CLINICAL TRIAL: NCT00779662
Title: The Prevalence of Rheumatic Heart Disease in School Children in Fiji
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Queensland Institute of Medical Research (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Menzies School of Health Research (Other); University of Melbourne (Other)
Responsible Party: Samantha Colquhoun, Menzies School of Health Research
Other Study IDs: 07- 0070; U01AI060579 (NIH)
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Rheumatic Heart Disease
Keywords: Rheumatic Heart Disease; Streptococcus; Fiji
MeSH Terms: conditions — Rheumatic Heart Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional

SUMMARY:
This study is an epidemiological observational cross-sectional study designed to estimate the prevalence of echocardiographically confirmed RHD in school children from 5-14 years of age in Fiji. The study will be conducted in the Central Division of Fiji within a selection of up to16 primary schools located in the Korovou/Tailevu and Rewa/Nausori sub-divisions. School children will be enrolled after informed consent has been obtained. A standard cardiac examination (auscultation) will be performed as part of the routine annual health check by both school nurses, who have attended a training workshop, and by a paediatrician. All children with or without murmur will have a screening echocardiogram performed at a subsequent visit. Children found to have possible, probable or definite RHD or other cardiac pathology on the screening echocardiogram, will have a full echocardiogram performed by the echocardiography technician at the time of the second study visit. They will all also be referred to a paediatric cardiologist for further investigation and management and monitoring . Cases of RHD will be referred to and followed up by the National Fiji RHD register based at CWMH in Suva.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will be obtained for all participants
* All children between the ages of 5-14 Years are eligible for the study.

Exclusion Criteria:

* None

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will be conducted in the Central Division of Fiji within a selection of up to16 primary schools located in the Korovou/Tailevu and Rewa/Nausori sub-divisions.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)